CLINICAL TRIAL: NCT01229124
Title: SCOR in Targeted Therapies for Infant Leukemias Project 4: MicroRNA Sequencing of Infant AML
Brief Title: RNA Biomarkers in Tissue Samples From Infants With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B1; COG-AAML11B1 (Other: Children's Oncology Group); NCI-2011-02841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Base Sequence; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: nucleic acid sequencing
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in RNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying RNA biomarkers in tissue samples from infants with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Sequence the microRNAs present in 20 infant AML samples as a pilot study.
* Compare microRNAs present in infant AML samples to infant ALL samples that are being concurrently sequenced in a separate study to identify lineage- and translocation-specific microRNAs.

OUTLINE: This is a multicenter study.

Previously collected cryopreserved cells from diagnosis are sequenced using reverse transcriptase-PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Available cryopreserved cells from diagnosis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosis of acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sequence of the microRNAs present in 20 infant acute myeloid leukemia (AML) samples
Comparison of microRNAs present in infant AML samples to infant acute lymphoblastic leukemia samples to identify lineage- and translocation-specific microRNAs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cleary, MD, Principal Investigator — Stanford University